CLINICAL TRIAL: NCT01947452
Title: The Effects of Summer Employment on Disadvantaged Youth: Experimental Evidence
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Chicago (Other)
Collaborators: City of Chicago Department of Family and Support Services (Unknown); Cook County Office of the President (Unknown); Walmart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB12-1112
Record Dates: First submitted 2012-08-17; First posted 2013-09-20 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-08

CONDITIONS: Reduce Violence and Crime; Increase School Engagement; Increase Future Labor Market Outcomes
Keywords: Youth violence reduction; Youth crime reduction; School engagement; Employment; Social-emotional learning
MeSH Terms: interventions — Employment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jobs Only (Experimental): Youth will be offered a 5-hour per day, 5-day per week employment opportunity over 7 weeks. They will be paid the Illinois minimum wage of $8.25 per hour.
  Interventions: Behavioral: Employment
- Jobs plus Social-Emotional Learning (Experimental): Youth will be offered a 3-hour per day, 5-day per week employment opportunity over 7 weeks. They will also be offered 2-hour per day, 5-day per week social-emotional learning programming, for which they will be paid the same hourly wage as their job ($8.25/hour).
  Interventions: Behavioral: Employment; Behavioral: Social-Emotional Learning

INTERVENTIONS:
Behavioral: Employment — Community organizations will place youth in summer jobs based on youth interests and the availability of positions. Jobs will be part-time in non-profit and government organizations. Youth will be paid the IL minimum wage of $8.25 per hour. The community organizations will provide job mentors to assist youth with barriers to work like transportation or clothing, and to provide supervision at the job site.
Behavioral: Social-Emotional Learning — Community organizations will provide 2 hours of social-emotional learning programming for 5 hours a day. The programming is based on cognitive behavioral therapy principles designed to help youth learn to understand and manage their emotions and behavior. It seeks to teach: self awareness (recognizing one's emotions and values as well as one's strengths and limitations), self management (managing emotions and behaviors to achieve one's goals), social awareness (showing understanding and empathy for others), relationship skills (forming positive relationships, working in teams, and dealing effectively with conflict), and responsible decision-making (making ethical, constructive choices about personal and social behavior).
  Arms: Jobs plus Social-Emotional Learning

SUMMARY:
Chicago's Department of Family and Support Services will be providing summer employment and social-emotional skill training to youth over the summer of 2012. The investigators are partnering with them to evaluate the effects of the program. The investigators will track applicants to the program through existing administrative databases to assess the short- and long-term effects of the government's program. The investigators hypothesize that the program will decrease violence involvement and criminal activity, increase schooling engagement, and increase future employment outcomes.

DETAILED DESCRIPTION:
The unemployment rates facing American youth are bleak. Youth employment over the summer, when teenagers are most likely to work, is at a 60 year low. The last decade has shown a dramatic drop: 44.1 percent of teens were employed in July 2000, but only 25.6 percent were working in July 2010. The situation for minority and low-income youth is even worse: the 2010 employment rate for low-income black teens in Illinois was less than one-fourth the rate for higher-income white teens (9 vs. 39 percent).

There are good reasons to think that this level of teen unemployment will create significant social costs as well as life-long consequences for youth. Teen employment has been shown to significantly increase employment outcomes later in life; one study from the late 1990s finds that working 20 hours a week as a high school senior increases earnings by 22 percent and wages by 10 percent 6-9 years later. Increasing wages for teens - both immediately through the provision of a job itself and later through increased earning potential - may also have a substantial impact on their crime rates. There is evidence that the higher the wage rate available to an individual, the less likely he is to commit a violent or property crime. Increasing income more generally (through income transfers, housing vouchers, tax credits, etc.) has also been convincingly shown to reduce crime, as has investing in individuals' skill development. Since the provision of a summer job is likely to perform all three functions - increase the available wage, provide additional income, and improve individuals' skills (not to mention keep youth busy during the summer months when crime usually spikes) - it is reasonable to expect that it would also decrease criminal behavior.

Surprisingly, there is almost no direct evidence on the effects of providing teens with summer jobs. Some early evaluations of programs in the 70s and 80s showed promising but mixed results, yet the research designs were too weak to draw strong conclusions. In addition, none of those evaluations looked at criminal behavior or violence involvement as outcomes, which seem likely to be one of the key effects of such programs. Less direct evidence shows that intensive residential job training programs have created substantial decreases in arrests, convictions, and incarceration for participants, and that job placement programs can reduce crime among parolees and increase incomes among welfare recipients. Taken together, the evidence suggests that using employment as a crime reduction strategy is quite promising, if not yet proven. But for summer jobs programs in particular, there is a startling lack of evidence.

Despite the dearth of research, policymakers already seem convinced that summer employment support is a good idea. The federal government dedicated $1.2 billion of the 2009 stimulus to employment for disadvantaged youth, with an emphasis on summer jobs programs. These spending levels are not new. Summer jobs for disadvantaged youth have been federally funded since 1964; from 1998 to the present, they have been part of the annual appropriation for Youth Activities of about $1 billion. The President proposed another $1.5 billion specifically for youth summer jobs last fall; when Congress did not pass his proposal, he committed the Department of Labor to arranging for 250,000 youth summer opportunities regardless.

Given the amount of resources spent on youth summer jobs programs over the past half century, the lack of evidence on such programs' effects is startling. Because of the way Chicago's jobs program for disadvantaged youth - One Summer +PLUS - is structured, the program will produce some of the only rigorous evidence to date on the effects of summer jobs programs. It will also measure the incremental effectiveness of adding a social-cognitive skill development component. Similar social-cognitive programming has been shown to reduce violent crime and increase school engagement in a recent randomized control trial. The evaluation will also assess the cost effectiveness of both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in one of 13 target high schools in Chicago, or
* Expecting to enroll in one of 13 target high schools for fall 2012
* Between ages 14 and 21 at program start

Exclusion Criteria:

* None

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1634 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Criminal activity | Program start through end of program (8 weeks)
  The number of each of four subtypes of arrests (violent, property, drug, and other) will be measured using individual-level administrative data on juvenile and adult arrests from the Chicago Policy Department.
Criminal activity | 6 months post-program
  The number of each of four subtypes of arrests (violent, property, drug, and other) will be measured using individual-level administrative data on juvenile and adult arrests from the Chicago Policy Department.
Criminal activity | 1 year post-program
  The number of each of four subtypes of arrests (violent, property, drug, and other) will be measured using individual-level administrative data on juvenile and adult arrests from the Chicago Policy Department.
Criminal activity | 18 months post-program
  The number of each of four subtypes of arrests (violent, property, drug, and other) will be measured using individual-level administrative data on juvenile and adult arrests from the Chicago Policy Department.
Criminal activity | 2 years post-program
  The number of each of four subtypes of arrests (violent, property, drug, and other) will be measured using individual-level administrative data on juvenile and adult arrests from the Chicago Policy Department.

SECONDARY OUTCOMES:
School engagement | 6 months after program start (Dec 2013)
  Schooling outcomes will be measured using student-level administrative data from the Chicago Public Schools. Engagement will be assessed using data on attendance, grades, course-taking, disciplinary incidents, test scores, graduation, school switching, and enrollment in schools within juvenile justice facilities.
School engagement | 1 year post-program start (June 2014)
  Schooling outcomes will be measured using student-level administrative data from the Chicago Public Schools. Engagement will be assessed using data on attendance, grades, course-taking, disciplinary incidents, test scores, graduation, school switching, and enrollment in schools within juvenile justice facilities.
School engagement | 18 months post-program start (Dec 2014)
  Schooling outcomes will be measured using student-level administrative data from the Chicago Public Schools. Engagement will be assessed using data on attendance, grades, course-taking, disciplinary incidents, test scores, graduation, school switching, and enrollment in schools within juvenile justice facilities.
School engagement | 2 years post-program start (June 2014)
  Schooling outcomes will be measured using student-level administrative data from the Chicago Public Schools. Engagement will be assessed using data on attendance, grades, course-taking, disciplinary incidents, test scores, graduation, school switching, and enrollment in schools within juvenile justice facilities.
Employment | 6 months post-program start
  Employment and wages will be measured using individual-level quarterly earnings records from Unemployment Insurance, provided by the Illinois Department of Employment Security.
Employment | 12 months post-program start
  Employment and wages will be measured using individual-level quarterly earnings records from Unemployment Insurance, provided by the Illinois Department of Employment Security.
Employment | 18 months post-program start
  Employment and wages will be measured using individual-level quarterly earnings records from Unemployment Insurance, provided by the Illinois Department of Employment Security.
Employment | 24 months post-program start
  Employment and wages will be measured using individual-level quarterly earnings records from Unemployment Insurance, provided by the Illinois Department of Employment Security.
Victimization | Program start through end of program (8 weeks)
  Number of victimization/incident reports in the Chicago Police Department victimization records (reports made to police by victims).
Victimization | 6 months post-program
  Number of victimization/incident reports in the Chicago Police Department victimization records (reports made to police by victims).
Victimization | 12 months post-program
  Number of victimization/incident reports in the Chicago Police Department victimization records (reports made to police by victims).
Victimization | 18 months post-program
  Number of victimization/incident reports in the Chicago Police Department victimization records (reports made to police by victims).
Victimization | 24 months post-program
  Number of victimization/incident reports in the Chicago Police Department victimization records (reports made to police by victims).

CONTACTS AND LOCATIONS:
Overall Officials: Harold Pollack, PhD, Principal Investigator — University of Chicago; Sara Heller, MPP, Study Director — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Bellotti J, Rosenberg L, Sattar S, Esposito AM, Ziegler J. Reinvesting in America's Youth: Lessons from the 2009 Recovery Act Summer Youth Employment Initiative. Mathematica Policy Research. Washington, D.C., 2010.
- [Background] Bloom D, Gardenire-Crooks A, Mandsager C. Reengaging high school dropouts: Early results of the National Guard ChalleNGe Program evaluation. MDRC report, 2009.
- [Background] Center for Labor Market Studies. The Depression in the Teen Labor Market in Illinois in Recent Years. Report, 2012.
- [Background] Fernandes-Alcantara, AL. Vulnerable Youth: Federal Funding for Summer Job Training and Employment. Congressional Research Service Report, 2011.
- [Background] Gould, ED, Weinberg BA, Mustard DB. Crime rates and local labor market opportunities in the United States: 1979-1997. The Review of Economics and Statistics 84(1): 45-61, 2002.
- [Background] Grogger, J. Market Wages and Youth Crime. Journal of Labor Economics 16(4), 756-791, 1998.
- [Background] Hamilton, G. Moving People from Welfare to Work: Lessons from the National Evaluation of Welfare-to-Work Strategies. MDRC Report, 2002.
- [Background] Heller S, Jacob BA, Ludwig J. Family Income, Neighborhood Poverty, and Crime. In Controlling Crime: Strategies and Tradeoffs, Eds. Philip J. Cook, Jens Ludwig and Justin McCrary. National Bureau of Economic Conference Report, University of Chicago Press, 2011.
- [Background] Hill, PL, Roberts BW, Grogger JT, Guryan J, Sixkiller K. Decreasing Delinquency, Criminal Behavior, and Recidivism by Intervening on Psychological Factors Other Than Cognitive Ability: A Review of the Intervention Literature. In Controlling Crime: Strategies and Tradeoffs,Eds. Philip J. Cook, Jens Ludwig and Justin McCrary. National Bureau of Economic Conference Report, University of Chicago Press: 367-406, 2011.
- [Background] Redcross C, Bloom D, Azurdia G, Zweig J, Pindus N. Implementation, Two-Year Impacts, and Costs of the Center for Employment Opportunities (CEO) Prisoner Reentry Program. MDRC Report, 2009.
- [Background] Ruhm, C. Is High School Employment Consumption or Investment? Journal of Labor Economics 15(4): 735-776, 1997.
- [Background] Schochet P, Burghardt J, McConnel S. Does Job Corps work? Impact findings from the National Job Corps Study. American Economic Review 98(5): 1864-86, 2008.
- [Background] Heller S, Pollack H, Ander R, Ludwig J. Improving Social-Cognitive Skills among Disadvantaged Youth: A Randomized Field Experiment. University of Chicago Working Paper, 2011.